CLINICAL TRIAL: NCT04440228
Title: Adapting and Implementing TeamSTEPPS in School Mental Health
Brief Title: TeamSTEPPS in School Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 834488
Record Dates: First submitted 2020-06-08; First posted 2020-06-19 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Child Behavior Problem; Multidisciplinary Communication; Interprofessional Relations
Keywords: school-based mental health; TeamSTEPPS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Schools implementing TeamSTEPPS (Experimental): Select schools will take a participatory approach to collaboratively identify solutions to challenges in collocated school-based mental health services based upon the feedback of stakeholders and use TeamSTEPPS to support mental health team-school collaboration.
  Interventions: Behavioral: TeamSTEPPS

INTERVENTIONS:
Behavioral: TeamSTEPPS — TeamSTEPPS is an evidence-based approach for teams that can be adapted for school mental health.
  Team Strategies and Tools to Enhance Performance and Patient Safety (TeamSTEPPS), has been widely disseminated in health care settings with promising outcomes. TeamSTEPPS is designed to build competencies in the areas of leadership, situation monitoring, mutual support, and communication and has been associated with improvements in teamwork and communication as well as patient outcomes, such as decreased seclusion in psychiatric hospitals.

SUMMARY:
Team Strategies and Tools to Enhance Performance and Patient Safety (TeamSTEPPS) is an evidence-based approach for teams that can be adapted for school mental health. TeamSTEPPS has been widely disseminated in health care settings with promising outcomes. TeamSTEPPS is designed to build competencies in the areas of leadership, situation monitoring, mutual support, and communication and has been associated with improvements in teamwork and communication as well as patient outcomes, such as decreased seclusion in psychiatric hospitals. This approach has yet to be extended as an implementation strategy in school or community mental health teams. If an evidence-based team approach like TeamSTEPPS can be successfully applied to school mental health teams, it could provide a cost-effective strategy for improving student mental health services and bolstering existing EBP implementation efforts, which to date generally have been insufficient in producing long-term clinician behavior change. In Aim 1 the investigators will capture key stakeholder perspectives about challenges in collocated school mental health services through formative work to inform collaborative planning and capacity building activities in Aim 2. Then, in Aim 2 the investigators will identify inter-organizational challenges and required components of TeamSTEPPS to adapt. The investigators will establish an advisory board and adapt TeamSTEPPS. The product of Aim 2 will be an adapted TeamSTEPPS, directed toward both school mental health and school-employed personnel, and specific, tailored implementation strategies to improve services in schools in conjunction with TeamSTEPPS. Finally, In Aim 3 the investigators will explore the feasibility, acceptability, and utility of TeamSTEPPS and the strategies generated in Aim 2 on inter-professional collaboration, teamwork, and student outcomes in eight schools.

ELIGIBILITY:
Inclusion Criteria:

* Must be one of the following: mental health providers, teachers, leaders from schools (e.g., principals), leaders from community mental health agencies (i.e., executive directors, clinical supervisors), and leadership personnel from the payer or partner school district.

Exclusion Criteria:

* There are no exclusion criteria proposed for school and agency-employed personnel. Participants will not be excluded given their gender, demographics, and/or past experience.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Benjamin Wolk, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make data from our trial available for other researchers by uploading it to the National Clinical Trials Database. The proposed research will include data from 95 school mental health providers, teachers, and administrators and supervisors overseeing school mental health services in Philadelphia public schools. The final dataset will include quantitative (socio-demographic characteristics, school characteristics, outcomes, and contextual predictors of implementation) data. We will collect identifiers required to create a Global Unique Identifier (GUID) that will allow for inclusions in the National Database of Clinical Trials. We also will include recommended language in our consent forms related to obtain participant permission to upload their data to the National Database.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The descriptive data will be uploaded every six months during data collection periods of the study. All other data will be submitted at time of the publication of the manuscripts describing our main findings.
Access Criteria: Any data directly shared with other investigators would entail a data-use agreement, signed by the research team, our system partners, and the individual(s) requesting data, and that accounts for (1) commitment to using the data only for research and as outlined and approved in the agreement; (2) IRB approval at the host institution, (3) a plan for securing the data using appropriate technology, and (4) an agreed upon plan to destroy or return the data upon completion. In such cases, we will make the data and associated documentation available to users under our own auspices, such as by sending an encrypted hard-drive to users.

REFERENCES:
- [Derived] Kuriyan A, Kinkler G, Cidav Z, Kang-Yi C, Eiraldi R, Salas E, Wolk CB. Team Strategies and Tools to Enhance Performance and Patient Safety (TeamSTEPPS) to Improve Collaboration in School Mental Health: Protocol for a Mixed Methods Hybrid Effectiveness-Implementation Study. JMIR Res Protoc. 2021 Feb 8;10(2):e26567. doi: 10.2196/26567. PMID 33555258

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were school staff recruited from school mental health teams working across three school districts.
Pre-assignment Details: Participants were existing employees working across three partner school districts. There was no randomization or assignment to study arms/conditions, though because participants naturally existed within the three districts, we report some analyses by district unit. All participants across all districts received the same intervention (i.e., TeamSTEPPS training).
Units Other Than Participants: School Districts
Groups:
- Schools Implementing TeamSTEPPS: We conducted a quasi-experimental, single-arm pilot study of an adapted TeamSTEPPS curriculum for school mental health team members. Team Strategies and Tools to Enhance Performance and Patient Safety (TeamSTEPPS), has been widely disseminated in health care settings with promising outcomes. TeamSTEPPS is designed to build competencies in the areas of leadership, situation monitoring, mutual support, and communication and has been associated with improvements in teamwork and communication as well as patient outcomes, such as decreased seclusion in psychiatric hospitals. All participants, who were employees working across three partner school districts, completed training in TeamSTEPPS, the primary intervention.
Period: Overall Study
Arm/Group | Schools Implementing TeamSTEPPS
Started | 90; 3 School Districts
Completed | 66; 3 School Districts
Not Completed | 24; 0 School Districts

BASELINE CHARACTERISTICS:
Groups:
- Schools Implementing TeamSTEPPS: We conducted a quasi-experimental, single-arm pilot study of an adapted TeamSTEPPS curriculum for school mental health team members. Team Strategies and Tools to Enhance Performance and Patient Safety (TeamSTEPPS) is designed to build competencies in the areas of leadership, situation monitoring, mutual support, and communication and has been associated with improvements in teamwork and communication as well as patient outcomes, such as decreased seclusion in psychiatric hospitals. All participants across all school districts received training in TeamSTEPPS which is the primary intervention in this trial.
Arm/Group | Schools Implementing TeamSTEPPS
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data was missing for one participant
  years
    number analyzed (Participants) | 89
    (all) | 38.73 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data were missing for two participants
  Participants
    number analyzed (Participants) | 88
    Female | 70
    Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 84
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 70
  More than one race | 1
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention Measure (FIM)
Description: Reliable and validated 4-item tool to assess perceptions of the feasibility of an intervention (in this case, TeamSTEPPS training). Each item may be scored 1 = "completely disagree", 2 = "disagree", 3 = "neither agree nor disagree", 4 = "agree", or 5 = "completely agree." An overall mean score (possible score range from 1 to 5) across the 4 items is computed, where higher scores indicate more positive perceptions of intervention feasibility.
Time Frame: assessed immediately post-training in TeamSTEPPS (on average, 4 hours after completion of baseline measures)
Population: Staff that completed TeamSTEPPS training
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Schools Implementing TeamSTEPPS: We conducted a quasi-experimental, single-arm pilot study of an adapted TeamSTEPPS curriculum for school mental health team members. Team Strategies and Tools to Enhance Performance and Patient Safety (TeamSTEPPS), has been widely disseminated in health care settings with promising outcomes. TeamSTEPPS is designed to build competencies in the areas of leadership, situation monitoring, mutual support, and communication and has been associated with improvements in teamwork and communication as well as patient outcomes, such as decreased seclusion in psychiatric hospitals.
Arm/Group | Schools Implementing TeamSTEPPS
Number analyzed (Participants) | 74
score on a scale | 4.25 (0.57)

2. Primary Outcome: Acceptability of Intervention Measure (AIM)
Description: Reliable and validated 4-item observational tool to assess perceptions of the acceptability of an intervention (in this case, TeamSTEPPS training). Each item may be scored 1 = "completely disagree", 2 = "disagree", 3 = "neither agree nor disagree", 4 = "agree", or 5 = "completely agree." An overall mean score (possible score range from 1 to 5) across the 4 items is computed, where higher scores indicate greater perceptions of intervention acceptability.
Time Frame: assessed immediately post-training in TeamSTEPPS (on average, 4 hours after completion of baseline measures)
Population: Staff that completed TeamSTEPPS training
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Schools Implementing TeamSTEPPS
Number analyzed (Participants) | 74
score on a scale | 4.28 (.68)

3. Secondary Outcome: Oxford Non-Technical Skills (NOTECHS) Scale
Description: Validated 4-item observational tool to assess teamwork and cognitive skills in teams. Items reflect team skills in leadership and management; teamwork and cooperation; problem-solving and decision making; and situational awareness. An observer codes team behavior in each domain using 3-5 items rated from 1 (Below Standard) to 4 (Excellent). An overall mean score, ranging from 1 to 4, is computed across items, where higher scores indicate stronger teamwork skills.
Time Frame: Assessed at baseline (i.e., on average, 1 week prior to training in TeamSTEPPS), immediately post-training in TeamSTEPPS (on average, 1 week after completion of baseline observation), and at 6- and 12-month follow-ups.
Population: Staff trained in TeamSTEPPS, observed in district teams. When multiple observations occurred by multiple raters at a time point, we computed mean (SD) ratings across raters.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: School Districts
Groups:
- Schools Participating in TeamSTEPPS: All participants, across schools, who completed training in TeamSTEPPS.
Arm/Group | Schools Participating in TeamSTEPPS
Number analyzed (Participants) | 90
Number analyzed (School Districts) | 3
units on a scale
  Baseline | 2.40 (0.33)
  Post-training | 3.33 (0.13)
  6 month follow-up | 3.38 (0.52)
  12 month follow-up | 2.88 (1.11)
Statistical Analysis 1: Comparison: Schools Participating in TeamSTEPPS; Repeated measures ANOVA examining change over time across the three partner school districts; Test type: Superiority; p = 0.088, ANOVA — Assumptions of ANOVA were violated, so we conducted a Related-Samples Friedman's Two-Way Analysis of Variance by Ranks; F=6.54, df=3

4. Other Pre Specified Outcome: Expanded School Mental Health Collaboration Instrument (ESMHCI)
Description: 59-item tool to assess perceptions of aspects of collaboration between school professionals and mental health professionals from collaborating agencies on a continuous scale. An average score is calculated, with higher scores indicating strengths and lower scores indicating areas to consider improving or targeting. Responses for all items on the scale are measured on one of two, four-point Likert-type scales (1 = never to 4 = often for items related to Types of Collaboration; and 1 = strongly disagree to 4 = strongly agree for items related to Influences on Collaboration and Perceived Benefits of Collaboration). A mean total score is computed, with possible scores ranging from 1 to 4, with higher scores indicating stronger collaboration.
Time Frame: Assessed at baseline (i.e., pre-training in TeamSTEPPS) and and at 6- and 12-month follow-ups. Six- and 12-month follow-up scores were averaged to create a single follow-up score.
Population: Staff that completed TeamSTEPPS training
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Schools Implementing TeamSTEPPS
Number analyzed (Participants) | 51
score on a scale
  Baseline | 2.83 (0.54)
  Follow-up | 3.01 (0.57)
Statistical Analysis 1: Comparison: Schools Implementing TeamSTEPPS; We conducted paired t-tests to evaluate simple pre-to-post changes in the primary outcome measures. We fitted linear mixed-effects regression models for each outcome variable, specifying random intercepts for participant ID to account for repeated measures and within-individual clustering. The core model included a binary post-training indicator as the primary predictor, along with the baseline value of the corresponding outcome as a covariate; Test type: Superiority; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 0.204, 95% CI 2-sided [0.036 to 0.373]

5. Other Pre Specified Outcome: TeamSTEPPS Teamwork Perceptions Questionnaire (T-TPQ)
Description: Self-report measure of individual perceptions of group-level team skills and behavior. It is based upon the five core components of teamwork that comprise TeamSTEPPS, totaling 35 items. Items are rated continuously on a five-point scale from strongly disagree = 1 to strongly agree = 5. A mean total score is computed by averaging all items (possible score range = 1 to 5). Higher scores indicate more favorable perceptions of teamwork.
Time Frame: Assessed at baseline (i.e., pre-training in TeamSTEPPS) and at 6- and 12-month follow-ups. Six- and 12-month follow-up scores were averaged to create a single follow-up score.
Population: Staff that completed TeamSTEPPS training
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Schools Implementing TeamSTEPPS
Number analyzed (Participants) | 57
score on a scale
  Baseline | 3.77 (0.51)
  Follow-Up | 3.76 (.55)
Statistical Analysis 1: Comparison: Schools Implementing TeamSTEPPS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .277, Regression, Linear; Mean Difference (Final Values) = 0.078, 95% CI 2-sided [-0.064 to 0.219]

6. Other Pre Specified Outcome: TeamSTEPPS Teamwork Attitudes Questionnaire (T-TAQ)
Description: Self-report measure of individual attitudes related to the core components of teamwork captured within TeamSTEPPS. Six items measure each of the core teamwork constructs, for a total of 30 items. Items are rated continuously on a five-point scale from strongly disagree = 1 to strongly agree = 5. A mean total score is calculated across items with a possible score range of 1 to 5. Higher scores indicated more positive attitudes toward teamwork.
Time Frame: as for outcome 5
Population: Staff that completed TeamSTEPPS training
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Schools Implementing TeamSTEPPS
Number analyzed (Participants) | 57
score on a scale
  Baseline | 4.43 (0.31)
  Follow-up | 4.42 (0.29)
Statistical Analysis 1: Comparison: Schools Implementing TeamSTEPPS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.996, Regression, Linear; Mean Difference (Final Values) = 0.002, 95% CI 2-sided [-0.082 to 0.083]

ADVERSE EVENTS:
Time Frame: Participants were enrolled, on average, for a 1 year period.
Arm/Group | Schools Implementing TeamSTEPPS
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT04440228/Prot_SAP_000.pdf